CLINICAL TRIAL: NCT00004915
Title: Phase II Study of Raloxifene in Recurrent Endometrial Cancer
Brief Title: Raloxifene in Treating Patients With Persistent or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 98G1; NU-98G1; NCI-G00-1710
Record Dates: First submitted 2000-03-07; First posted 2004-08-30 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Endometrial Cancer
Keywords: recurrent endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: raloxifene

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of endometrial cancer cells. Hormone therapy using raloxifene may fight endometrial cancer by reducing the production of estrogen.

PURPOSE: Phase II trial to study the effectiveness of raloxifene in treating patients who have persistent or recurrent endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine response rate and time to disease progression in patients with recurrent endometrial cancer treated with raloxifene. II. Determine overall survival in these patients treated with this regimen. III. Determine the toxicity of raloxifene in this patient population.

OUTLINE: Patients receive oral raloxifene daily. Treatment continues indefinitely in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 13-50 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Recurrent endometrial cancer Evidence of persistent or recurrent disease 4 weeks following primary treatment with radiation and surgery Bidimensionally measurable disease Not a candidate for curative salvage radiotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No history of unexplained or uncontrolled thromboembolic disease No active thromboembolic disease Other: No active or uncontrolled second malignancy HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy for early stage or advanced endometrial cancer Endocrine therapy: At least 4 weeks since prior hormonal therapy for early stage or advanced endometrial cancer Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-11; Primary Completion 2000-02 (Actual); Study Completion 2000-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Y. Roland, MD, Study Chair — Florida Gynecologic Oncology - Fort Myers
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States